CLINICAL TRIAL: NCT02337322
Title: Immune Reconstitution in Severely Immunosuppressed Antiretroviral-naive HIV-1-Infected Patients (<100 CD4+ T Cells/μL) Taking Antiretroviral Regimens Based on Dolutegravir or Ritonavir-boosted Darunavir (the Advanz-4 Trial).
Brief Title: Immune Recovery in Advanced , ARV-naïve, HIV-1-infected Individuals Taking Dolutegravir or Ritonavir-boosted Darunavir
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Juan A. Arnaiz (Other)
Responsible Party: Sponsor-Investigator, Juan A. Arnaiz, MD, PhD, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Advanz-4
Record Dates: First submitted 2015-01-09; First posted 2015-01-13 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Acquired Immune Deficiency Syndrome Virus
Keywords: Acquired Immune Deficiency Syndrome Virus; HIV; HIV-1; Antiretroviral treatment; HIV Advanced Disease; AIDS; Dolutegravir; Darunavir
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABC+3TC+DTG (Active Comparator): Abacavir+lamivudine+Dolutegravir, QD, Single tablet Regimen
  Interventions: Drug: Dolutegravir
- ABC+3TC+DRV/r (Active Comparator): Abacavir+lamivudine+ritonavir-boosted darunavir, QD
  Interventions: Drug: Darunavir/r

INTERVENTIONS:
Drug: Dolutegravir
  Arms: ABC+3TC+DTG
Drug: Darunavir/r
  Other Names: Ritonavir-boosted Darunavir
  Arms: ABC+3TC+DRV/r

SUMMARY:
There are few randomized clinical trials in advanced HIV patients. This is a multicenter, randomized, open clinical trial, comparing 2 parallel groups, to compare the immunological reconstitution and the virological efficacy and safety of 2 different combinations of antiretroviral therapy given once a day (QD): abacavir plus lamivudine plus either dolutegravir, or darunavir-ritonavir during 96 weeks in advanced antiretroviral naïve HIV-1 infected patients with less than 100 CD4+ T-cells/mm3. Primary endpoint is the median increase in CD4+ T-cell count at 48 weeks after starting HAART.

ELIGIBILITY:
Inclusion Criteria:

1. HIV patients > 18 years old who provide signed and dated informed consent.
2. Male and female.
3. Chronic HIV infection.
4. Antiretroviral naïve.
5. Confirmed CD4+ T cell count below 100 cells/mm3
6. HLA B5701 negative patients.

Exclusion Criteria:

1. Active opportunistic infections requiring parenteral treatment
2. Patients with cryptococcal meningitis treated with voriconazole
3. AIDS-defining cancers needing chemotherapy.
4. Female patients pregnant or breastfeeding.
5. Patients with documented history of allergy to sulfonamides.
6. Any contraindications to study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Median CD4 T cell count increase | 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic of Barcelona, Barcelona, BCN, Spain

REFERENCES:
- [Derived] Miro JM, Torres F, Manzardo C, Bonfill E, Curran A, Domingo P, Podzamczer D, Paredes R, Force L, Falco V, Gutierrez M, Saumoy M, Castelli A, Inciarte A, Rovira C, Cruceta A, Hurtado C, Climent N, Lozano F, Plana M; Advanz-4 investigators. Immune reconstitution in very advanced HIV patients treated with dolutegravir vs. darunavir-based triple antiretroviral therapy: the Advanz-4 randomized clinical trial. Clin Microbiol Infect. 2026 Jan;32(1):169-176. doi: 10.1016/j.cmi.2025.09.026. Epub 2025 Oct 11. PMID 41083105